CLINICAL TRIAL: NCT00167349
Title: Cardiopulmonary Bypass and Inflammatory Response
Acronym: CPB-I
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: John A. Kellum, MD, University of Pittsburgh School of Medicine
Other Study IDs: 0306088
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Thoracic Surgery; Cardiopulmonary Bypass
Keywords: cardiac surgery; cardiopulmonary bypass; cytokines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if a difference exists in the inflammatory response which occurs related to coronary artery bypass graft (CABG)surgery performed on cardiopulmonary bypass as compared to CABG surgery performed off bypass at the University of Pittsburgh Medical Center.

DETAILED DESCRIPTION:
Acute inflammatory response occurring in cardiopulmonary bypass (CPB) patients has been clearly associated with deleterious clinical outcomes. Increasing understanding of the pathophysiology of systemic inflammatory response syndrome (SIRS) following CPB has facilitated the development of strategies to attenuate the damaging effects of cytokine-induced inflammation. For any strategy to be tested, one needs to clearly define and understand the inflammatory response occurring with CPB. Although this has been extensively studied, there is wide variation in the reported time course and magnitude of this response. This variation is, in part, due to the heterogeneous nature of the patient population studied (variable severity of illnesses, ejection fractions, co-morbidities, etc.). Hence, in our study, we propose to study the inflammatory response occurring in patients undergoing coronary artery bypass graft (CABG) with and without the use of CPB in our institution, and to determine whether the severity of inflammatory response seen in CABG patients is associated with impairment of any specific clinical parameter in the immediate post-operative period (i.e., ventricular dysfunction, lung injury, bleeding, renal failure, etc).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing CABG and/or patients undergoing other procedures (i.e., valve surgery, myomectomy, etc.) in addition to coronary revascularization
* Age: 18 years up to and including 90 years

Exclusion Criteria:

* Patient is not scheduled to undergo CABG surgery
* Ejection Fraction £ 30%
* Chronic renal failure requiring hemodialysis
* Long-term steroid use prior to surgery
* HIV positive patients (HIV testing will not be required to rule out HIV)
* Status post organ transplantation or on immune modulating drugs
* Presence of severe sepsis in the past month prior to surgery
* Prisoners

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CABG patients
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2003-12; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Kellum, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Rimmele T, Venkataraman R, Madden NJ, Elder MM, Wei LM, Pellegrini RV, Kellum JA. Comparison of inflammatory response during on-pump and off-pump coronary artery bypass surgery. Int J Artif Organs. 2010 Mar;33(3):131-8. doi: 10.1177/039139881003300301. PMID 20383854